CLINICAL TRIAL: NCT02669693
Title: Effect of Olives on Glycaemic Response in Vivo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Gary Williamson, Professor, University of Leeds
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MEEC 12-037a
Record Dates: First submitted 2016-01-19; First posted 2016-02-01 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Diabetes
Keywords: Olives, oleuropein
MeSH Terms: conditions — Diabetes Mellitus | interventions — Bread

ARMS (2):
- bread without olives (Placebo Comparator): Intervention (no olives): Subjects will consume a meal of 109 g white bread and 200 of ml water, and post-prandial blood glucose measured over a 3 hour period.
  Interventions: Dietary Supplement: bread without olives
- bread with olives (Active Comparator): Intervention (olives 100 g): Subjects will consume a meal of 109 g white bread, 100 g of olives and 200 of ml water, and post-prandial blood glucose measured over a 3 hour period.
  Interventions: Dietary Supplement: bread with olives

INTERVENTIONS:
Dietary Supplement: bread without olives
  Arms: bread without olives
Dietary Supplement: bread with olives
  Arms: bread with olives

SUMMARY:
This research is aimed at determining whether the presence of oleuropein in olives (Olea europaea L.) has any lowering effect on post-prandial blood glucose levels. Volunteers will be required to consume commercially available olives together with white bread, and their glycaemic response will be measured. The blood glucose response of bread will be determined initially as a control/reference. Food samples and control will be consumed in random order.

The recent rise in the cases of Diabetes mellitus in both children and adults has raised a concern for the need to proffer immediate solutions amongst scientists in the fields of medicine food science and nutrition. One of the approaches of reducing postprandial hyperglycaemia and high glucose spikes is to impede digestion and absorption of starch. This is potentially achieved through the inhibition of the activities of starch digesting enzymes namely alpha amylase and alpha glycosidase. There are currently some antidiabetic drugs such as acarbose and miglitol which have been quite efficient in these inhibitory functions but not without associated side effects and complications such as liver toxicity, etc, arising from to long term usage of such drugs. It therefore becomes imperative for natural substitutes from food sources to be explored as better alternatives. At the moment several plant foods are under investigation as suitable alternatives, and olives appear to be quite promising in this regard. There are quite a few studies that have reported the inhibitory activities of olives oleuropein on alpha amylase in vitro but information on in vivo testing is very scarce.

It is expected that the research outcome will be a gateway to the reduction and control of the incidence of diabetes mellitus.

DETAILED DESCRIPTION:
Prior to commencement of the study, potential volunteers will be given a clear, concise Participant Information Sheet and Informed Consent Form by the investigator to read, complete and sign in their own time. The investigator will answer all questions to the satisfaction of the individual and will not influence the decision of taking part in the study. The participants will be free to withdraw from the study at any point without providing a reason. The written consent form will be signed and dated at least 2 days prior to enrolment in the study by the volunteers and the Investigator. It will be photocopied and one copy will be kept by the Investigator (for the study records) and one by the volunteer. Participation by the volunteers is conditional upon receiving the written consent by the volunteer.

Candidates will be asked to complete a questionnaire in order to assess their suitability for the study. The information pertains to their lifestyle and may be considered a sensitive issue, however each volunteer will be assured of confidentiality and that participation is entirely voluntary. The information on the questionnaire will include height, weight, gender, age and relevant medical history. Confidentiality of all participants' information will be maintained. Identification will be coded using random ID numbers that will be assigned on the day of study. All data collected will be treated as confidential and stored securely in a locked filing cabinet according to current University regulations. The linkage between individual identity and ID number will be kept in written form only and stored in a locked filling cabinet in a restricted access area, thus it will not be possible to identify individual participants from the ID numbers. Data evaluation will only be performed using ID numbers. In accordance with the University guidelines on the password protected M-drive of the University server, anonymised data will be stored for at least 5 years.

Blood glucose will be measured after consumption of test meal/control using a commercially available glucometer which is available to be bought by any member of the public and people already use them on their own. It measures glucose concentrations immediately and meets the accuracy requirement for the ISO 15197 standard. A drop of blood is enough and is obtained from participants by means of a mild finger prick using a sterile puncture device designed for this purpose for each time point. The finger prick protocol is the WHO/FAO 1998 glycaemic index approved protocol. Nine (9) finger pricks will be needed (0, 15, 30, 45, 60, 90, 120, 150 and 180minutes) will be needed per study session.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75
* Fasting glucose (blood glucose level before breakfast) 3.9 -5.9mmol/L

Exclusion Criteria:(self assessed)

* Diabetic
* on long term prescribed medication (except contraceptives)
* pregnant or lactating
* on special diet (for losing weight or fruit extracts supplements)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Post-prandial blood glucose concentration | 180 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Gary Williamson, PhD, Principal Investigator — University of Leeds
Locations (1):
- School of Food Science and Nutrition, University of Leeds, Leeds, West Yorkshire, United Kingdom